CLINICAL TRIAL: NCT00794443
Title: A Multi-center Double-blind Parallel-group Comparison Study in Involutional Osteoporosis Patients to Examine the Efficacy and Safety of ONO-5920/YM529 Monthly Intermittent Formulation With Its Daily Formulation.
Brief Title: ONO-5920/YM529 Confirmatory Study in Involutional Osteoporosis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 529-CL-028; ONO-5920-05
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Osteoporosis; Bone Loss, Age-Related
Keywords: ONO-5920; YM529; Bone mineral density; Minodronic acid
MeSH Terms: conditions — Osteoporosis | interventions — YM 529

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1. Monthly - Dose 1 (Experimental): Monthly intermittent administration, dose 1
  Interventions: Drug: YM529 / ONO-5920
- 2. Monthly - Dose 2 (Experimental): Monthly intermittent administration, dose 2
  Interventions: Drug: YM529 / ONO-5920
- 3. Daily (Active Comparator): Daily administration
  Interventions: Drug: YM529 / ONO-5920

INTERVENTIONS:
Drug: YM529 / ONO-5920 — Oral
  Other Names: YM529; ONO-5920; Minodronic acid

SUMMARY:
This is a multi-center double-blind parallel-group study in involutional osteoporosis patients to compare the efficacy and safety of monthly oral intermittent formulation ONO-5920/YM529 with its daily formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose bone mineral density is <70% of Young Adult Mean (YAM), or <80% of YAM who have fragile fracture history
* Patients can walk on his/her own
* Written informed consent has been obtained from the patient.

Exclusion Criteria:

* Sequential osteoporosis patients or patients with other disorders showing low bone mass
* Patients with the findings that influence measurement of lumbar vertebral bone mineral density by the DXA method
* Patients who are unable to keep raising or standing for ≥30 min
* Patients with peptic ulcer
* Patients who have experienced anamnesis or gastrectomy (total extraction)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Percent changes in the lumbar vertebral bone mineral density (L2-4BMD) by the DXA method | At the final evaluation point

SECONDARY OUTCOMES:
Time-course changes in the percent change of bone metabolism markers | Through the treatment period
Time-course changes in the total femoral bone mineral density by the DXA method | Through the treatment period
Assessment of adverse events, lab test values | Through the treatment period
Frequency of fracture | At the final evaluation point

CONTACTS AND LOCATIONS:
Overall Officials: Toshiomi Minamide, Study Director — Ono Pharmaceutical Co. Ltd; Central Contact, Study Chair — Clinical Development Administration Dept., Astellas Pharma Inc.
Locations (5):
- Japan (5):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Shikoku